CLINICAL TRIAL: NCT05051098
Title: The European HBV Registry: a Joint Initiative of TherVacB and DZIF
Brief Title: A Non-interventional Registry for Patients with Hepatitis B Virus Infection
Status: Recruiting | Type: Observational
Sponsor: Hannover Medical School (Other)
Collaborators: European Union (Other); German Center for Infection Research (Other); German Liver Foundation (DLS) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3374-2016; 848223 (Other Grant/Funding Number: European Union); 05.220 (Other Grant/Funding Number: German Center for Infection Research (DZIF))
Record Dates: First submitted 2021-08-25; First posted 2021-09-21 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Hepatitis B Virus Infection
MeSH Terms: conditions — Hepatitis B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- TherVacB Subgroup: No interventions. The participating study centers of the EU funded project "TherVacB" recruit patients with stricter inclusion- and exclusion criteria, hence forming a sub-cohort.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
In order to tackle the unmet needs in chronic HBV infection, a consortium of clinical partners has gathered to establish a registry for patients with hepatitis B mono- and co-infections. The partners will build up a European-wide registry to be able to stratify patients for upcoming clinical trials.

Extensive analyses of virus and host-specific parameters are to be carried out from these patients. The knowledge gained thereby should contribute to a better understanding of the HBV control and enable patient stratification with regard to immunomodulatory therapies.

Furthermore, hepatitis B patients are to be identified who are willing to participate in future studies to investigate immunotherapies to cure HBV infections (e.g. therapeutic vaccines).

ELIGIBILITY:
Inclusion Criteria:

* Hepatitis B Virus Infection

TherVacB sub-cohort:

* confirmed chronic hepatitis B virus infection: HBsAg positive for at least 1 year prior inclusion
* HBeAg status documented for at least 6 months

Exclusion Criteria:

TherVacB sub-cohort:

* age >70 years
* co-infection with HIV, HCV (RNA positive),
* clinically relevant concomitant liver diseases (ALD, NASH, Haemochromatosis, Autoimmune hepatitis, AT1, Wilson's disease, primary biliary cirrhosis etc.)
* significant comorbidities (e.g. malignancies)
* immunosuppressive treatment (> 40 mg Cortisol- equivalent)
* liver cirrhosis (judged clinically or based on ultrasound/transient elastography)
* History of hepatocellular carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in day clinic or outpatient clinic at the participating study centers.
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2021-05-06 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with change HBsAg levels | 5 years
  Regular assessment of quantitative HBsAg levels
Number of patients with seroconversion to anti-HBs | 5 years
  Measurement of quantitative HBsAg and anti-HBs levels
Quantification of IL6, IP-10, IFNg and IL1beta and correlation with HBsAg and ALT levels | 5 years
  Cytokine and Chemokine quantification in patients for subsequent correlation with viral parameters

SECONDARY OUTCOMES:
Number of patients with hepatitis B related increased or decreased quality of life | 5 years
  Regular assessment of QOL by SF36 questionnaires.
Number of patients with hepatitis B related HCC (hepatocellular carcinoma) | 5 years
  Regular assessment of HCC status
Number of patients with hepatitis B related liver cirrhosis | 5 years
  Regular assessment of liver status
Number of patients with hepatitis B related death | 5 years
  Regular quantification of lost-to-follow-up reasons.

CONTACTS AND LOCATIONS:
Overall Officials: Markus Cornberg, Principal Investigator — Hannover Medical School; Xavier Forns, Principal Investigator — Fundacio Clinic per a la Recerca Biomedica
Locations (1):
- Hannover Medical School, Hanover, Germany

IPD SHARING:
Plan to Share IPD: Undecided
Undecided which and where data will be shared. Depends on regulatory requirements of EU and German Federal Ministry of Education and Research

REFERENCES:
- See also: Website of the EU funded part of the registry — https://www.thervacb.eu/patients/the-european-hbv-patient-registry/